CLINICAL TRIAL: NCT06599606
Title: Investigation of the Relationship Between Ultrasonographic Muscle Thickness Measurement and Echogenicity Assessment with Functional Scales in Patients with Spinal Muscular Atrophy: an Observational, Cross-Sectional, Case-Control Study
Brief Title: Ultrasonographic Muscle Assessment and Functional Scales in Spinal Muscular Atrophy
Status: Active, not recruiting | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Eren Aygun, Medical Doctor, Istanbul University - Cerrahpasa
Other Study IDs: IstanbulUC-EAygun-01
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Spinal Muscular Atrophy (SMA); Neuromuscular Disease
Keywords: Spinal Muscular Atrophy (SMA); Muscle Ultrasonography; Muscle Thickness; Functional Scales; Disease Progression; Objective Biomarkers
MeSH Terms: conditions — Muscular Atrophy, Spinal; Neuromuscular Diseases; Disease Progression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Case: Patients diagnosed with spinal muscular atrophy (SMA) who have received at least four loading doses of nusinersen
  Interventions: Diagnostic Test: Ultrasonographic Assessment
- Control: Healthy, age- and sex-matched control individuals
  Interventions: Diagnostic Test: Ultrasonographic Assessment

INTERVENTIONS:
Diagnostic Test: Ultrasonographic Assessment — A researcher will perform all ultrasonographic measurements using the ESAOTE My Lab 70 model ultrasound device with a 4-13 MHz linear probe. System settings will be kept constant throughout each study, and all images will be obtained using this single ultrasound device. Only the depth will be adjusted to optimally assess the relevant muscle. The muscle thickness measurement protocol with ultrasound includes four muscles on the dominant side of each child: two proximal upper and lower extremity muscles (biceps brachii/brachialis and quadriceps) and two distal upper and lower extremity muscles (forearm flexors and tibialis anterior). In the assessment of muscle echogenicity, images will be transferred to ImageJ software to calculate luminance ratios (LR).

SUMMARY:
This study aims to investigate the relationship between ultrasonographic muscle thickness measurement and echogenicity assessment with functional scales in children with spinal muscular atrophy (SMA). By utilizing ultrasonographic techniques, the study seeks to provide objective biomarkers for assessing muscle health and monitoring treatment response. Currently, the evaluation of SMA often relies on subjective clinical assessments; this study addresses that gap by offering more precise and objective indicators of disease progression and functional status. The ultimate goal is to improve treatment strategies and enhance patient outcomes through better assessment tools.

DETAILED DESCRIPTION:
Spinal muscular atrophy (SMA) is a neuromuscular disorder that typically leads to progressive lower motor neuron loss from early childhood. The most common form is caused by deletions in the survival motor neuron 1 (SMN1) gene, inherited in an autosomal recessive manner. SMA is classified into at least three subtypes based on the age of onset and the level of motor development achieved. In Type 1 SMA (severe form), symptoms usually appear before 6 months of age, and children are unable to sit unsupported. In Type 2 SMA (intermediate form), symptoms start between 6 and 18 months, and children cannot walk unsupported. Type 3 SMA (mild form) presents after the second year of life, and affected children can walk unsupported. Although the exact prevalence and carrier rates of SMA in our country are not fully determined, it is estimated that there are between 130 and 180 new cases annually, given approximately 1,200,000 live births each year. The total number of SMA patients in the country is about 3,000.

Despite current treatments, muscle weakness and significant functional loss affecting quality of life are commonly observed in SMA patients. At present, the efficacy of SMA treatment is measured through clinical assessment, including monitoring of changes in motor developmental milestones and functional scales. However, the lack of objective biomarkers that are less reliant on patient cooperation, as opposed to functional scales, complicates monitoring treatment response for patients. Establishing reliable methods to assess disease progression and treatment response is crucial for conducting robust clinical studies.

Musculoskeletal ultrasonography presents itself as a suitable imaging modality for use as a biomarker in SMA management due to its non-invasiveness, repeatability, absence of radiation, ability to evaluate multiple muscles quickly, and ease of application. Furthermore, the feasibility of performing ultrasonographic examinations at the bedside facilitates access to a larger number of patients, especially those with limited mobility or requiring respiratory support. Previous literature has reported the advantages of muscle ultrasonography in evaluating neuromuscular disorders, including SMA.

In conclusion, this study, which will investigate the relationship between ultrasonographic muscle thickness measurement and echogenicity evaluation and functional scales in patients diagnosed with SMA for the first time in our country, will guide physicians and researchers seeking to assess disease progression, determine treatment efficacy, and develop rehabilitation strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age between 0-18 years
* Confirmed diagnosis of SMA through genetic testing
* Having received four loading doses of nusinersen
* Written consent provided for participation in the study

Exclusion Criteria:

* History of surgical operation or trauma in the muscles to be examined
* Presence of spasticity that complicates positioning of the extremities and hinders ultrasound imaging

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients diagnosed with spinal muscular atrophy (SMA) who are being followed at the Department of Pediatric Neurology and the Department of Physical Medicine and Rehabilitation at Cerrahpaşa Medical Faculty
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Muscle Thickness Measurement | Baseline
  Muscle thickness in specific muscle groups will be assessed using ultrasonography. Measurements will include biceps brachii/brachialis, quadriceps, forearm flexors, and tibialis anterior. Thickness will be measured at predetermined anatomical sites using electronic calipers.
Muscle Echogenicity Assessment | Baseline
  Muscle echogenicity will be assessed by calculating luminance ratios (LR) from ultrasonographic images. Luminance ratios will be calculated for the target muscle groups (biceps brachii/brachialis, quadriceps, forearm flexors, tibialis anterior, triceps, proximal hamstrings, gastrosoleus) and compared to subcutaneous tissue. This will involve measuring and analyzing images using ImageJ software.

SECONDARY OUTCOMES:
CHOP-INTEND | Baseline
  CHOP-INTEND (Childrens Hospital of Philadelphia Infant Test of Neuromuscular Disorders) is a clinical scale designed to assess the motor function of infants with type 1 SMA or other types of SMA who cannot sit unsupported. This scale comprises 16 items that focus on evaluating the infant's movements, posture, and reflexes.
HFMSE | Baseline
  HFMSE (Hammersmith Functional Motor Scale-Expanded) is a scale used to assess motor skills in patients with type 2 and type 3 SMA who can sit unsupported. It consists of 33 items that score various movements, including sitting, rolling in a prone position, lifting the head in a prone position, rising, kneeling, standing, walking, jumping, and climbing stairs.
RULM | Baseline
  RULM (Revised Upper Limb Module) is a scale designed to assess functional abilities in the upper extremities of SMA patients. The scale includes an entry item to determine functional levels and consists of 19 items covering both distal and proximal movements.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University - Cerrahpasa (IUC), Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hodgkinson VL, Oskoui M, Lounsberry J, M'Dahoma S, Butler E, Campbell C, MacKenzie A, McMillan HJ, Simard L, Vajsar J, Brais B, Chapman KM, Chrestian N, Crone M, Dobrowolski P, Dojeiji S, Dowling JJ, Dupre N, Genge A, Gonorazky H, Hasal S, Izenberg A, Johnston W, Leung E, Lochmuller H, Mah JK, Marerro A, Massie R, McAdam L, McCormick A, Melanson M, Mezei MM, Nguyen CE, O'Connell C, O'Ferrall EK, Pfeffer G, Phan C, Plamondon S, Poulin C, Rodrigue X, Schellenberg KL, Selby K, Sheriko J, Shoesmith C, Smith G, Taillon M, Taylor S, Warman Chardon J, Worley S, Korngut L. A National Spinal Muscular Atrophy Registry for Real-World Evidence. Can J Neurol Sci. 2020 Nov;47(6):810-815. doi: 10.1017/cjn.2020.111. Epub 2020 Jun 4. PMID 32493524
- [Background] Nakamura R, Kitamura A, Tsukamoto T, Otowa Y, Okamoto N, Ogawa N, Yamakawa I, Kim H, Sanada M, Urushitani M. Spinal Muscular Atrophy Type 3 Showing a Specific Pattern of Selective Vulnerability on Muscle Ultrasound. Intern Med. 2021 Jun 15;60(12):1935-1939. doi: 10.2169/internalmedicine.6396-20. Epub 2021 Jan 15. PMID 33456041
- [Background] Coratti G, Carmela Pera M, Montes J, Scoto M, Pasternak A, Bovis F, Sframeli M, D'Amico A, Pane M, Albamonte E, Antonaci L, Lia Frongia A, Mizzoni I, Sansone VA, Russo M, Bruno C, Baranello G, Messina S, Dunaway Young S, Glanzman AM, Duong T, de Sanctis R, Stacy Mazzone E, Milev E, Rohwer A, Civitello M, Darras BT, Bertini E, Day J, Muntoni F, De Vivo DC, Finkel RS, Mercuri E. Revised upper limb module in type II and III spinal muscular atrophy: 24-month changes. Neuromuscul Disord. 2022 Jan;32(1):36-42. doi: 10.1016/j.nmd.2021.10.009. Epub 2021 Nov 7. PMID 34980538
- [Background] Moreira AL, Mendonca RH, Polido GJ, Oliveira MCB, Silva AMS, Zanoteli E. Muscle Ultrasound Changes Correlate With Functional Impairment in Spinal Muscular Atrophy. Ultrasound Med Biol. 2023 Jul;49(7):1569-1574. doi: 10.1016/j.ultrasmedbio.2023.02.021. Epub 2023 Apr 8. PMID 37037685
- [Background] Ng KW, Connolly AM, Zaidman CM. Quantitative muscle ultrasound measures rapid declines over time in children with SMA type 1. J Neurol Sci. 2015 Nov 15;358(1-2):178-82. doi: 10.1016/j.jns.2015.08.1532. Epub 2015 Aug 28. PMID 26432577
- [Background] Wu JS, Darras BT, Rutkove SB. Assessing spinal muscular atrophy with quantitative ultrasound. Neurology. 2010 Aug 10;75(6):526-31. doi: 10.1212/WNL.0b013e3181eccf8f. PMID 20697104
- [Background] Abraham A, Drory VE, Fainmesser Y, Algom AA, Lovblom LE, Bril V. Muscle thickness measured by ultrasound is reduced in neuromuscular disorders and correlates with clinical and electrophysiological findings. Muscle Nerve. 2019 Dec;60(6):687-692. doi: 10.1002/mus.26693. Epub 2019 Sep 10. PMID 31478199
- [Background] Mah JK, van Alfen N. Neuromuscular Ultrasound: Clinical Applications and Diagnostic Values. Can J Neurol Sci. 2018 Nov;45(6):605-619. doi: 10.1017/cjn.2018.314. PMID 30430964
- [Background] Heckmatt JZ, Pier N, Dubowitz V. Real-time ultrasound imaging of muscles. Muscle Nerve. 1988 Jan;11(1):56-65. doi: 10.1002/mus.880110110. PMID 3277050
- [Background] Pillen S, Arts IM, Zwarts MJ. Muscle ultrasound in neuromuscular disorders. Muscle Nerve. 2008 Jun;37(6):679-93. doi: 10.1002/mus.21015. PMID 18506712
- [Background] Antonaci L, Pera MC, Mercuri E. New therapies for spinal muscular atrophy: where we stand and what is next. Eur J Pediatr. 2023 Jul;182(7):2935-2942. doi: 10.1007/s00431-023-04883-8. Epub 2023 Apr 17. PMID 37067602
- [Background] Pane M, Palermo C, Messina S, Sansone VA, Bruno C, Catteruccia M, Sframeli M, Albamonte E, Pedemonte M, D'Amico A, Brigati G, de Sanctis R, Coratti G, Lucibello S, Bertini E, Vita G, Danilo Tiziano F, Mercuri E; Italian EAP Working Group. An observational study of functional abilities in infants, children, and adults with type 1 SMA. Neurology. 2018 Aug 21;91(8):e696-e703. doi: 10.1212/WNL.0000000000006050. Epub 2018 Jul 25. PMID 30045959
- [Background] De Sanctis R, Coratti G, Pasternak A, Montes J, Pane M, Mazzone ES, Young SD, Salazar R, Quigley J, Pera MC, Antonaci L, Lapenta L, Glanzman AM, Tiziano D, Muntoni F, Darras BT, De Vivo DC, Finkel R, Mercuri E. Developmental milestones in type I spinal muscular atrophy. Neuromuscul Disord. 2016 Nov;26(11):754-759. doi: 10.1016/j.nmd.2016.10.002. Epub 2016 Oct 5. PMID 27769560
- [Background] Chabanon A, Seferian AM, Daron A, Pereon Y, Cances C, Vuillerot C, De Waele L, Cuisset JM, Laugel V, Schara U, Gidaro T, Gilabert S, Hogrel JY, Baudin PY, Carlier P, Fournier E, Lowes LP, Hellbach N, Seabrook T, Toledano E, Annoussamy M, Servais L; NatHis-SMA study group. Prospective and longitudinal natural history study of patients with Type 2 and 3 spinal muscular atrophy: Baseline data NatHis-SMA study. PLoS One. 2018 Jul 26;13(7):e0201004. doi: 10.1371/journal.pone.0201004. eCollection 2018. PMID 30048507
- [Background] Kolb SJ, Kissel JT. Spinal Muscular Atrophy. Neurol Clin. 2015 Nov;33(4):831-46. doi: 10.1016/j.ncl.2015.07.004. PMID 26515624